CLINICAL TRIAL: NCT00127452
Title: Alpha Omega Trial: A Randomised, Placebo Controlled, Double Blind Intervention Study of the Effect of Low Doses of Omega-3 Fatty Acids on Cardiovascular Diseases in Patients With a History of Myocardial Infarction
Brief Title: Alpha Omega Trial: Study of Omega-3 Fatty Acids and Coronary Mortality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Netherlands Heart Foundation (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Unilever R&D (Industry)
Responsible Party: Daan Kromhout, Wageningen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: METC-ZWH 0552; NHF-2000T401; L01.049; 5R01HL076200 (NIH); NCT00139464 (obsolete NCT alias)
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Cardiovascular Diseases
Keywords: alpha-linolenic acid; cardiovascular diseases; coronary heart disease; coronary patients; DHA; dietary intervention; dietary supplementation; docosahexaenoic acid; eicosapentaenoic acid; EPA; fish oil; fish fatty acids; human subjects; ischaemic heart disease; margarine; marine fatty acids; mortality; myocardial infarction; n-3 fatty acids; n-3 polyunsaturated fatty acids; n-3 PUFA; omega-3 fatty acids; omega-3 polyunsaturated fatty acids; prevention; randomized controlled trial; secondary prevention
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- EPA + DHA (Experimental): Margarine spread that yields 400 mg of eicosapentaenoic acid (EPA) + docosahexaenoic acid (DHA) per day for average margarine use of 20 grams per day
  Interventions: Dietary Supplement: margarine spread
- ALA (Experimental): Margarine spread that yields 2 grams of alpha-linolenic acid (ALA) per day for average margarine use of 20 grams per day
  Interventions: Dietary Supplement: margarine spread
- EPA + DHA plus ALA (Experimental): Margarine spread that yields 400 mg of EPA + DHA per day plus 2 grams of ALA per day, for average margarine use of 20 grams per day
  Interventions: Dietary Supplement: margarine spread
- Placebo (Placebo Comparator): Margarine spread that contains no EPA, DHA or ALA (exchanged for oleic acid)
  Interventions: Dietary Supplement: margarine spread

INTERVENTIONS:
Dietary Supplement: margarine spread — Daily use of margarine spread (approximately 20 grams) during 40 months

SUMMARY:
The Alpha Omega Trial is a randomized, placebo-controlled, double-blind dietary intervention study in 4837 postmyocardial infarction patients in the Netherlands to examine whether incidence of cardiovascular diseases during 40 months of follow-up can be prevented by low doses of omega-3 polyunsaturated fatty acids. The key objectives are:

* to examine the effect of low-dose supplementation (400 mg/day) of eicosapentaenoic acid and docosahexaenoic acid on incidence of cardiovascular diseases; and
* to examine the effect of low-dose supplementation (2 g/day) of alpha-linolenic acid on incidence of cardiovascular diseases.

DETAILED DESCRIPTION:
Whether dietary omega-3 (or n-3) polyunsaturated fatty acids are causally related to risk of cardiovascular diseases (CVD) is a major, unresolved question in preventive cardiology. Essential n-3 fatty acids are eicosapentaenoic acid (EPA; C20:5, n-3) and docosahexaenoic acid (DHA; C22:6, n-3) on one hand, and their parent compound alpha-linolenic acid (ALA; C18:3, n-3) on the other hand. The intake of n-3 fatty acids is below recommended levels in most Western populations. The Alpha Omega Trial is a randomized, double-blind, placebo-controlled study of the effect of low-dose supplementation of ALA and EPA-DHA on CVD. A total of 4837 Dutch men and women aged 60-80 years who had a myocardial infarction in the past 10 years are randomly allocated to 2 g/d of ALA, 400 mg/d of EPA-DHA, 2 g/d ALA + 400 mg/d EPA-DHA, or placebo, for 40 months. Increased intake of n-3 fatty acids is achieved through daily use of 20 g of margarine on bread. Margarines for all treatment groups are similar in taste and appearance. The primary outcome of the trial is 'major cardiovascular events', which comprises incident CVD and cardiac interventions (PCI and CABG) during follow-up. Secondary endpoints are incident CVD, fatal CVD, fatal CHD and all-causes mortality. Complete follow-up for vital status is achieved. Cause-specific mortality is coded by an independent Endpoint Adjudication Committee. Physical examination, blood sampling and data collection on diet and lifestyle are performed in all subjects at baseline, in 810 randomly selected subjects after 20 months of intervention, and in 58% of the cohort at the end of follow-up. Cardiovascular health, serious adverse events, lifestyle, fish intake and margarine use are monitored in all subjects by yearly telephone interviews. Compliance is continuously monitored by registration of margarine tubs. An objective biomarker of compliance (i.e. plasma n-3 fatty acids) is obtained in randomly selected subjects at baseline and after 20 and 40 months of intervention. The Alpha Omega Trial could provide a sound scientific basis for dietary recommendations on intake of ALA and EPA-DHA, in order to reduce the burden of cardiovascular diseases.

ELIGIBILITY:
Inclusion criteria:

* Men and women
* Aged 60 through 80 y
* Verified clinically diagnosed myocardial infarction up to 10 y before randomization
* Written informed consent

Exclusion criteria:

* Living in a nursing home or other institution
* Participation in another scientific study
* Habitual margarine intake < 10 g per day
* Habitual fish intake > 150 g per day
* Habitual alcohol intake > 6 drinks per day
* Use of fish oil capsules or other supplements containing omega-3 fatty acids
* Presence of cancer with < 1 y of life expectancy
* Cognitive impairment, as indicated by the Mini Mental State Examination (score <= 21)
* Unintended weight loss > 5 kg in the past year
* Lack of facilities for cooled margarine storage at home
* Inability or unwillingness to comply with study procedures

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4837 (Actual)
Dates: Start 2002-04; Primary Completion 2009-11 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Major cardiovascular events, which comprises fatal cardiovascular diseases (CVD), non-fatal myocardial infarction, non-fatal cardiac arrest, non-fatal stroke and cardiac interventions (PCI and CABG) | monitored during intervention

SECONDARY OUTCOMES:
Incident CVD, which comprises fatal CVD, non-fatal myocardial infarction, non-fatal cardiac arrest and non-fatal stroke | monitored during intervention
Fatal CVD, which comprises mortality from ischaemic heart disease, fatal cardiac arrest, sudden death undefined, mortality from heart failure and fatal stroke | monitored during intervention
Fatal CHD, which comprises mortality from ischaemic heart disease, mortality from cardiac arrest, and sudden death undefined | monitored during intervention
All-causes mortality | monitored during intervention
The composite of sudden death undefined and nonfatal and fatal cardiac arrest | monitored during intervention
The composite of sudden death undefined, nonfatal and fatal cardiac arrest, and self-reported placement of any implantable cardioverter-defibrillator, verified in medical records | monitored during intervention

CONTACTS AND LOCATIONS:
Overall Officials: Daan Kromhout, PhD MPH, Principal Investigator — Wageningen University, The Netherlands
Locations (32):
- Netherlands (32):
  - Medisch Centrum Alkmaar, Alkmaar
  - Flevo Ziekenhuis, Almere Stad
  - Meander Medisch Centrum, Amersfoort
  - Sint Lucas Andreas Ziekenhuis, Amsterdam
  - BovenIJ Ziekenhuis, Amsterdam
  - Slotervaartziekenhuis, Amsterdam
  - Gelre ziekenhuizen, Apeldoorn
  - Lievensberg Ziekenhuis, Bergen op Zoom
  - Rode Kruis Ziekenhuis, Beverwijk
  - IJsselland Ziekenhuis, Capelle aan den IJssel
  - Ziekenhuis Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - St. Anna Ziekenhuis, Geldrop
  - Oosterscheldeziekenhuis, Goes
  - Ziekenhuis Hilversum, Hilversum
  - Diaconessenhuis, Leiden
  - Rijnland Ziekenhuis, Leiderdorp
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Erasmus MC, Rotterdam
  - Havenziekenhuis, Rotterdam
  - Haga Ziekenhuis, location Leyweg, The Hague
  - Bronovo Ziekenhuis, The Hague
  - Haga Ziekenhuis, location Sportlaan, The Hague
  - Twee Steden Ziekenhuis, Tilburg
  - Maxima Medisch Centrum, Veldhoven
  - Alysis Ziekenhuis, Velp
  - Wageningen University, Division of Human Nutrition, Wageningen
  - Zaans Medisch Centrum, Zaandam
  - 't Lange Land ziekenhuis, Zoetermeer
  - Isala Klinieken, Zwolle

REFERENCES:
- [Background] Geleijnse JM, Giltay EJ, Schouten EG, de Goede J, Oude Griep LM, Teitsma-Jansen AM, Katan MB, Kromhout D; Alpha Omega Trial Group. Effect of low doses of n-3 fatty acids on cardiovascular diseases in 4,837 post-myocardial infarction patients: design and baseline characteristics of the Alpha Omega Trial. Am Heart J. 2010 Apr;159(4):539-546.e2. doi: 10.1016/j.ahj.2009.12.033. PMID 20362710
- [Derived] Liu S, Soedamah-Muthu SS, van Meerten SC, Kromhout D, Geleijnse JM, Giltay EJ. Use of benzodiazepine and Z-drugs and mortality in older adults after myocardial infarction. Int J Geriatr Psychiatry. 2023 Jan;38(1):e5861. doi: 10.1002/gps.5861. PMID 36514248
- [Derived] Pertiwi K, Wanders AJ, Harbers MC, Kupers LK, Soedamah-Muthu SS, de Goede J, Zock PL, Geleijnse JM. Plasma and Dietary Linoleic Acid and 3-Year Risk of Type 2 Diabetes After Myocardial Infarction: A Prospective Analysis in the Alpha Omega Cohort. Diabetes Care. 2020 Feb;43(2):358-365. doi: 10.2337/dc19-1483. Epub 2019 Nov 14. PMID 31727685
- [Derived] Sijtsma FP, Soedamah-Muthu SS, de Goede J, Oude Griep LM, Geleijnse JM, Giltay EJ, de Boer MJ, Jacobs DR Jr, Kromhout D. Healthy eating and lower mortality risk in a large cohort of cardiac patients who received state-of-the-art drug treatment. Am J Clin Nutr. 2015 Dec;102(6):1527-33. doi: 10.3945/ajcn.115.112276. Epub 2015 Oct 21. PMID 26490494
- [Derived] Hoogeveen EK, Geleijnse JM, Kromhout D, Stijnen T, Gemen EF, Kusters R, Giltay EJ. Effect of omega-3 fatty acids on kidney function after myocardial infarction: the Alpha Omega Trial. Clin J Am Soc Nephrol. 2014 Oct 7;9(10):1676-83. doi: 10.2215/CJN.10441013. Epub 2014 Aug 7. PMID 25104273
- [Derived] Hoogeveen EK, Geleijnse JM, Kromhout D, van't Sant P, Gemen EF, Kusters R, Giltay EJ. No effect of n-3 fatty acids supplementation on NT-proBNP after myocardial infarction: the Alpha Omega Trial. Eur J Prev Cardiol. 2015 May;22(5):648-55. doi: 10.1177/2047487314536694. Epub 2014 May 30. PMID 24879357
- [Derived] Brouwer IA, Geleijnse JM, Klaasen VM, Smit LA, Giltay EJ, de Goede J, Heijboer AC, Kromhout D, Katan MB. Effect of alpha linolenic acid supplementation on serum prostate specific antigen (PSA): results from the alpha omega trial. PLoS One. 2013 Dec 11;8(12):e81519. doi: 10.1371/journal.pone.0081519. eCollection 2013. PMID 24349086
- [Derived] Hoogeveen EK, Geleijnse JM, Kromhout D, Giltay EJ. No effect of n-3 fatty acids on high-sensitivity C-reactive protein after myocardial infarction: the Alpha Omega Trial. Eur J Prev Cardiol. 2014 Nov;21(11):1429-36. doi: 10.1177/2047487313494295. Epub 2013 Jun 17. PMID 23774275
- [Derived] Eussen SR, Geleijnse JM, Giltay EJ, Rompelberg CJ, Klungel OH, Kromhout D. Effects of n-3 fatty acids on major cardiovascular events in statin users and non-users with a history of myocardial infarction. Eur Heart J. 2012 Jul;33(13):1582-8. doi: 10.1093/eurheartj/ehr499. Epub 2012 Feb 1. PMID 22301766
- [Derived] Kromhout D, Geleijnse JM, de Goede J, Oude Griep LM, Mulder BJ, de Boer MJ, Deckers JW, Boersma E, Zock PL, Giltay EJ. n-3 fatty acids, ventricular arrhythmia-related events, and fatal myocardial infarction in postmyocardial infarction patients with diabetes. Diabetes Care. 2011 Dec;34(12):2515-20. doi: 10.2337/dc11-0896. PMID 22110169
- [Derived] Giltay EJ, Geleijnse JM, Kromhout D. Effects of n-3 fatty acids on depressive symptoms and dispositional optimism after myocardial infarction. Am J Clin Nutr. 2011 Dec;94(6):1442-50. doi: 10.3945/ajcn.111.018259. Epub 2011 Oct 26. PMID 22030221
- [Derived] Geleijnse JM, Giltay EJ, Kromhout D. Effects of n-3 fatty acids on cognitive decline: a randomized, double-blind, placebo-controlled trial in stable myocardial infarction patients. Alzheimers Dement. 2012 Jul;8(4):278-87. doi: 10.1016/j.jalz.2011.06.002. Epub 2011 Oct 2. PMID 21967845
- [Derived] Kromhout D, Giltay EJ, Geleijnse JM; Alpha Omega Trial Group. n-3 fatty acids and cardiovascular events after myocardial infarction. N Engl J Med. 2010 Nov 18;363(21):2015-26. doi: 10.1056/NEJMoa1003603. Epub 2010 Aug 28. PMID 20929341
- See also: Information site of the Alpha Omega Trial; statistical analysis plans are posted here — http://www.alphaomegatrial.com
- See also: Wageningen University and Research Centre — http://www.wur.nl
- See also: The Graduate School VLAG, Wageningen, The Netherlands — http://www.vlaggraduateschool.nl/
- See also: Netherlands Heart Foundation — http://www.hartstichting.nl